CLINICAL TRIAL: NCT04252976
Title: Meditation Based Lifestyle Modification in Healthy Individuals
Acronym: MBLM-H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonie Kliniken Zschadraß (Other)
Collaborators: Chemnitz University of Technology (Other)
Responsible Party: Principal Investigator, Holger C. Bringmann, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MBLM-H
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Mantra Meditation; Mantra Meditation + Body-Oriented Yoga; Mantra Meditation + Ethical Living; Mantra Meditation + Body-Oriented Yoga + Ethical Living

STUDY DESIGN:
Intervention Model Description: * 4 Treatment Conditions:
  * Multiple-baseline design: 3 Baselines (7, 14, 21 days)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mantra Meditation (Experimental): 8 weeks of mantra meditation with weekly group sessions.
  Interventions: Behavioral: Mantra Meditation
- Mantra Meditation plus Ethical Practice (Experimental): 8 weeks of mantra meditation plus ethical practice with weekly group sessions.
  Interventions: Behavioral: Ethical Living; Behavioral: Mantra Meditation
- Mantra Meditation plus Yoga Exercises (Experimental): 8 weeks of mantra meditation plus Yoga Exercises with weekly group sessions.
  Interventions: Behavioral: Yoga Exercises; Behavioral: Mantra Meditation
- Mantra Meditation plus Yoga Exercises plus Ethical Practice (Experimental): 8 weeks of mantra meditation plus Yoga Exercises plus ethical practice with weekly group sessions.
  Interventions: Behavioral: Ethical Living; Behavioral: Yoga Exercises; Behavioral: Mantra Meditation

INTERVENTIONS:
Behavioral: Ethical Living — Ethical principles based on Yoga philosophy, including contents of Yamas and Niyamas.
  Arms: Mantra Meditation plus Ethical Practice; Mantra Meditation plus Yoga Exercises plus Ethical Practice
Behavioral: Yoga Exercises — Ujjaii breathing and simple yoga asanas
  Arms: Mantra Meditation plus Yoga Exercises; Mantra Meditation plus Yoga Exercises plus Ethical Practice
Behavioral: Mantra Meditation — Meditation with mantras

SUMMARY:
MBLM is a holistic therapy for people with mental disorders whose positive effects on patients with depression have already been demonstrated in clinical use and a pilot study. In the present study, the differential effects of MBLM domains (ethical living, healthy lifestyle, and mantra meditation) on healthy volunteers will be investigated.

DETAILED DESCRIPTION:
MBLM expands existing concepts of mind-body medicine with ethical and spiritual concepts from the traditional Patanjali yoga system, which can act as a coping factor on the one hand, and higher motivation and deepening of practice (physical yoga exercises / mantra Meditation). MBLM aims to establish an exercise routine in the daily lives of the participants, which leads to salutogenesis. The promotion of mental health through meditation and yoga has been well documented (Büssing et al., 2012, Sedlmeier, Ebert, & Schwarz, 2012), also in clinical populations (Ospina et al., 2007). The preventive potential of the MBLM program will be examined for healthy volunteers, analogous to the already well-researched and widely used Mindfulness Based Stress Reduction program.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent

Exclusion Criteria:

1. Psychiatric disorder
2. Current participation in another meditation or yoga study
3. Regular existing meditation or yoga practice (more than once a week in the last 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change of Well-Being | Change from baseline Well-Being at 8 Weeks
  WHO (Five) Well-Being Index (WHO-5)
Change of Mind-Wandering | Change from baseline Mind-Wandering at 8 Weeks
  Mind Wandering Questionnaire
Change of Emotion regulation | Change from baseline Emotion Regulation at 8 Weeks
  Difficulties in Emotion Regulation Scale (DERS)
Change of Perceived Stress | Change from baseline Stress at 8 Weeks
  Perceived Stress Scale (PSS)
Change of Attention | Change from baseline Attention at 8 Weeks
  Sustained Attention to Response Task
Change of Body Awareness | Change from baseline body awareness at 8 Weeks
  Body Awareness Questionnaire
Life Satisfaction | Change from baseline life satisfaction at 8 Weeks
  Satisfaction with Life Scale
Course satisfaction | After 8 weeks of intervention
  Client Satisfaction Questionnaire
Adverse Events | After 8 weeks of intervention
  70 possible adverse events or extraordinary experiences associated with meditation or yoga practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Diakoniekliniken Zschadraß, Colditz, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
All data will be made available for free online access.
Supporting Information: Analytic Code
Time Frame: 2021

REFERENCES:
- [Derived] Matko K, Sedlmeier P, Bringmann HC. Differential Effects of Ethical Education, Physical Hatha Yoga, and Mantra Meditation on Well-Being and Stress in Healthy Participants-An Experimental Single-Case Study. Front Psychol. 2021 Aug 5;12:672301. doi: 10.3389/fpsyg.2021.672301. eCollection 2021. PMID 34421729